CLINICAL TRIAL: NCT01684787
Title: Open Multicentre, Phase IV Study to Evaluate Efficacy and Safety of Pegylated Interferon Alpha-2a (40 KD) Plus Ribavirin for Chronic Hepatitis C With Normal Transaminases in Human Immunodeficiency Virus-infected Patients
Brief Title: Study to Evaluate the Treatment for Chronic Hepatitis C With Normal Transaminases in HIV Positive Patients
Acronym: CONTRA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Miguel Santin (Other)
Responsible Party: Sponsor-Investigator, Miguel Santin, Dr, Hospital Universitari de Bellvitge
Organization: Hospital Universitari de Bellvitge (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Miguel Santín
Record Dates: First submitted 2010-06-11; First posted 2012-09-13 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-09

CONDITIONS: Chronic Hepatitis C
Keywords: chronic hepatitis C; normal ALT; HIV/HCV patients
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Peginterferon alfa-2a + ribavirin in normal ALT
  Interventions: Drug: Peginterferon alfa-2a + ribavirin in normal ALT
- 2 (Active Comparator): peginterferon alfa-2a + ribavirin in elevated ALT
  Interventions: Drug: Peginterferon alfa-2a + ribavirin in elevated ALT

INTERVENTIONS:
Drug: Peginterferon alfa-2a + ribavirin in normal ALT — peginterferon alfa-2a 180 mcg/weekly ribavirin 1000-1200 mg/daily
  Other Names: Pegasys + ribavirin
  Arms: 1
Drug: Peginterferon alfa-2a + ribavirin in elevated ALT — peginterferon alfa-2a 180 mcg/weekly ribavirin 1000-1200 mg/daily
  Other Names: Pegasys + ribavirin
  Arms: 2

SUMMARY:
In the current practice patients with normal levels of ALT were not treated. However, a percentage of patients will present an advanced grade of fibrosis and cirrhosis.

Another reason to treat is the similar response to the treatment than elevated ALT patients published recently in mono-infected patients.

The investigators have not data concerning the evolution and response to the treatment in co-infected patients with normal ALT.

In the story of treatment chronic hepatitis C of co-infected patients HCV/HIV, sometimes, it assumes a behavior similar between mono and co-infected patients and the results are different.

In the case of normal ALT the investigators do not know if the natural history in co-infected patients is similar than the mono-infected patients, and also the response of the treatment.

This study prospective and controls is the answer of this question. The main hypothesis is if the response of treatment in co-infected patients is not inferior than mono-infected patients.

The objective is to evaluate the efficacy and safety of peginterferon alfa-2a and ribavirin in HIV positive patients with chronic hepatitis and persistently normal ALT. Every CASE (patient with normal ALT) will have a CONTROL (patient with elevated ALT), concerning genotype, gender and hospital.

DETAILED DESCRIPTION:
The treatment of co-infected patients with normal ALT would be very important because the evolution of cirrhosis in this patients is quicker and frequently than mono-infected patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Hepatitis C co infected with stable HIV-1 and normal ALT (CASE) or elevated levels of ALT (CONTROL)
* CD4 > 200 cel/mL
* Stable anti-retroviral treatment for HIV during at least, the 6 previous months to the inclusion
* Negative contraception test
* Informed consent signed

Exclusion Criteria:

* Pregnancy
* Any previous treatment for CHC
* Any experimental treatment in the 6 previous weeks to the inclusion
* Cirrhosis grade B or C (Child-Pugh)
* Treatment with colony-stimulating factors, didanosine or zidovudine, immunomodulator therapy, isoniazid, rifampicin, …
* Hepatic cancer
* Neutrophils < 1500 cel/mL, Platelets < 70000 cel/mL, Hemoglobin < 11 g/dL (men) or < 12 g/dL (women) previous to inclusion
* Severe psychiatric illness background
* Serum creatinin > 1,5 times the upper normal limit
* Background of Pulmonary or Cardiovascular disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-09; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
% patients with RNA-HCV negative | 24 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Santin, Dr, Study Chair — Hospital Universitari of Bellvitge
Locations (18):
- Spain (18):
  - Hospital de Txagorritxu, Vitoria-Gasteiz, Alava
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Clinic, Barcelona, Barcelona
  - Consorci Sanitari Integral, Hospitalet, Barcelona
  - Hospital Universitari of Bellvitge, Hospitalet, Barcelona
  - Hospital General de Mataró, Mataró, Barcelona
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Hospital de Donostia, San Sebastián, Guipúzcoa
  - Hospital San Jorge, Huesca, Huesca
  - Hospital de la Princesa, Madrid, Madrid
  - Hospital Ramón y Cajal, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital 12 de Octubre, Madrid, Madrid
  - Hospital Xeral-Cíes, Vigo, Pontevedra
  - Hospital Joan XXIII, Tarragona, Tarragona
  - Hospital de Cruces, Barakaldo, Vizcaya
  - Hospital Clínico Lozano Blesa, Zaragoza, Zaragoza